CLINICAL TRIAL: NCT04201080
Title: A Phase 1, Two-part, Single Dose, Randomised, Double-blind, Placebo-controlled Parallel Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Subcutaneous TRV250 Following Glyceryl Trinitrate Infusion
Brief Title: A Trial to Evaluate the Efficacy, Safety and Tolerability of Subcutaneous TRV250
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because there have been significant enrollment struggles which has been exacerbated by the COVID impact. This has caused an undue delay to the study timelines and its enrollment goals beyond the business needs.
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CP250-1002
Record Dates: First submitted 2019-12-05; First posted 2019-12-17 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Migraines
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts: Part A is a proof of concept study; and Part B will be a dose ranging study
Who Masked: Participant, Investigator
Masking Description: Patients will be randomised to receive TRV250 20 mg or placebo in Part A and 1 of 3 doses of TRV250 or placebo in Part B. The study will be conducted in a double-blinded fashion (Investigator- and patient -blinded). Only unblinded personnel will have access to the randomisation list before official unblinding of treatment assignment. Interim analyses will be conducted at the end of Part A of the study prior to proceeding to Part B and the preliminary efficacy pharmacokinetic, safety and tolerability data will be evaluated unblinded at the end of Part A and shared with the Investigators in an unblinded manner, prior to starting Part B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: TRV250 for SC injection (Experimental): 2 SC injections of (10 mg/ml per injection)
  Interventions: Drug: Part A: TRV250-20mg/ml
- Part A: Placebo for SC injection (Placebo Comparator): 2 SC injections (identical to the TRV250)
  Interventions: Drug: Placebo
- Part B: TRV250 dose 1 for SC injection (Experimental): 1 of 3 doses of TRV250 (using 2 identical syringes)
  Interventions: Drug: Part B: TRV250 Dose 1
- Part B: TRV250 dose 2 for SC injection (Experimental): 1 of 3 doses of TRV250 (using 2 identical syringes)
  Interventions: Drug: Part B: TRV250 Dose 2
- Part B: TRV250 dose 3 for SC injection (Experimental): 1 of 3 doses of TRV250 (using 2 identical syringes)
  Interventions: Drug: Part B: TRV250 Dose 3
- Part B: Placebo for SC injection (Placebo Comparator): Placebo (using syringes identical to the TRV250 arms)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Part A: TRV250-20mg/ml — TRV250 SC Injections
  Other Names: Proof of concept
  Arms: Part A: TRV250 for SC injection
Drug: Placebo — Placebo SC injections
  Other Names: Proof of concept
  Arms: Part A: Placebo for SC injection
Drug: Part B: TRV250 Dose 1 — Dose 1of3 TRV250
  Other Names: Dose-ranging
  Arms: Part B: TRV250 dose 1 for SC injection
Drug: Part B: TRV250 Dose 2 — Dose 2of3 TRV250 SC injections
  Other Names: Dose-ranging
  Arms: Part B: TRV250 dose 2 for SC injection
Drug: Part B: TRV250 Dose 3 — Dose 3of3 TRV250 SC injections
  Other Names: Dose-ranging
  Arms: Part B: TRV250 dose 3 for SC injection
Drug: Placebo — Placebo SC injections
  Other Names: Dose-ranging
  Arms: Part B: Placebo for SC injection

SUMMARY:
A trial to assess the efficacy, safety, tolerability and effect of a drug (code name TRV250) given as an injection to subjects who have received an injection of a drug called glyceryl trinitrate (GTN) which is clinically known to induce an immediate headache of short duration (under 30 minutes), known as the "GTN immediate headache"

DETAILED DESCRIPTION:
This is a Phase 1, two-part, single dose, randomised, double-blind, placebo-controlled parallel study to evaluate the efficacy, safety, tolerability and pharmacokinetics of subcutaneous TRV250 following glyceryl trinitrate infusion-evoked migraine type headache.

Approximately 360 patients (120 in Part A and 240 in Part B) are planned to complete dosing and assessments.

Part A will be a proof of concept study; approximately 120 patients will be randomised to 1 of 2 treatments (60 patients per treatment arm). Patients will receive either TRV250 (20 mg) or placebo administered subcutaneously in a double-blind manner. Part B will be a dose-ranging study; approximately 240 patients will be randomised to 1 of 4 treatments (60 patients per treatment arm). Patients will receive 1 of 3 doses of TRV250 or placebo administered subcutaneously in a double-blind manner.

The study will consist of 3 phases: Screening, Confinement, and Follow-Up. Patients will participate in an outpatient Screening visit, a 3-day inpatient Confinement Phase that comprises GTN-infusion and treatment with TRV250 or placebo, and an outpatient safety Follow-Up visit 5 to 7 days post-dose.

The expected duration of participation is up to 6 weeks.

The diagnosis and criteria for inclusion covers male and female patients aged 18-55 years (inclusive), with a body mass index (BMI) within the range 18-32 kg/m2 inclusive at Screening. The patient must experience a migraine without aura as defined by International Headache Society (IHS) criteria 1.1 and experience between 1 migraine attack every other month to 8 migraine attacks per month. They should have had a positive outcome with Triptans, for their migraine attacks (Triptan Responders).

The investigational product (TRV250) will be administered by subcutaneous injection (10 mg/ml per injection). In Part A, 2 injections will be administered to deliver a single dose of 20 mg. In Part B, the dose levels to be administered will be decided following interim analysis of the data collected in Part A; however, the doses selected will not exceed that administered in Part A (up to 2 injections will be administered to deliver a single dose of up to 20 mg). Matched placebo injections will be administered by subcutaneous injections to maintain blinding.

By virtue of this being an exploratory study for the purpose of estimation and prediction, Bayesian estimates along with posterior predictive probabilities will be provided to address the primary and secondary efficacy objectives, as appropriate. Standard descriptive statistics will be provided to assess secondary safety and pharmacokinetic objectives.

Interim analyses will be conducted at the end of Part A of the study prior to proceeding to Part B. Preliminary pharmacokinetics (using nominal times) will be conducted to estimate the AUCt, AUC∞, Cmax, and t1/2. These preliminary efficacy, pharmacokinetic, safety and tolerability data will be evaluated unblinded at the end of Part A and shared with the Investigators in an unblinded manner, prior to starting Part B.

Once the study is complete, pharmacokinetic analyses will be completed using actual collection times.

In Part A, the difference in treatment proportions of patients who experience a headache occurring up to 4 hours post-dose will be tested using a chi-square. If the patient requires rescue medication then the patient will be considered a non-responder. In Part B, a Bayesian approach will be utilized using the prior information obtain from Part A. The proportion of patients who experience a headache occurring up to 4 hours post-dose, will be modelled using a Bayesian hierarchical logistic regression. This logistic regression will include a continuous covariate for TRV250 dose where Placebo is considered to be 0 mg of TRV250. If the patient requires rescue medication then the patient will be considered a non-responder.

Demographic and baseline data will be listed and summarised descriptively. Safety and tolerability assessments will be listed and summarised descriptively by treatment group as the observations and when appropriate, as the change from baseline. Plasma PK parameter values will be listed and summarised by treatment group. Dose proportionality may be assessed with a power model and slope analysis.

Safety laboratory tests will be tabulated and any out of range values highlighted. Clinically significant changes in safety laboratory results will be recorded as AEs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, aged between 18 and 55 years inclusive.
* Patient's Body Mass Index (BMI) is between 18 and 32 kg/m2 inclusive.
* Patient should have a clinical diagnosis of migraine without aura (IHS criteria 1.1) and experience between 1 migraine attack every other month to 8 migraine attacks per month. They should have had a positive outcome with Triptans, for their migraine attacks (Triptan Responders).

Exclusion Criteria:

* Patient has previous exposure to TRV250.
* Abnormal EEG at screening or risk factors of increased seizure potential, such as previous seizures, history of febrile seizures, cerebral tumor, stroke, cerebrovascular disease, or significant traumatic brain injury.
* Patient with a history of hypotension or hypertension, including where this is currently under control.
* Patient taking prophylactic migraine treatments such as beta blockers 28 days before GTN infusion on Day 1.
* Resting heart rate <45 beats per minute on assessment of vital signs at screening or pre-GTN infusion on Day 1.
* QTcF >450 msec at screening (mean of three ECGs) or pre-GTN infusion on Day 1.
* Patient with another headache disorder such as menstrual migraine, chronic migraine, cluster headache, tension headache or other chronic headache states.
* Patient who have a history, or family history of any vascular intracranial lesion such as subarachnoid aneurysm or similar and patients with a relevant neurological history.
* Patients who have any allergies/contraindications for Triptan administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is the proportion of patients who experienced a headache from dosing up to 4 hours post-dose, that exceeds a verbal numerical rating scale (NRS) headache rating of ≥2 points. | 0-4 hours post-dose
  Verbal Numerical Rating (NRS) and Headache Characteristics (Pain Response, Pain Freedom, Nausea, Photophobia) Assessment: 0 minutes prestart of GTN infusion and every 15 minutes until 4 hours post-dose

SECONDARY OUTCOMES:
The proportion of patients who experienced a headache occurring at various timepoints from dosing up to 8 hours post-dose, that exceeds a verbal NRS headache rating of ≥2 points | 0-8 hours post-dose
  NRS Headache Rating and Characteristics: 0 Minutes (mins) pre-start of GTN, every 15mins to 4 hours (hrs) post-dose, every 30mins to 8hrs post-dose
The proportion of patients who experience a headache occurring at various timepoints from dosing up to 8 hours post-dose, that exceeds a verbal NRS headache rating of ≥3 points. | 0-8 hours post-dose
  NRS Headache Rating and Characteristics: 0 Minutes (mins) pre-start of GTN, every 15mins to 4 hours (hrs) post-dose, every 30mins to 8hrs post-dose
The proportion of patients who experience a headache occurring at various timepoints from dosing up to 8 hours post-dose, that exceeds a verbal NRS headache rating of ≥4 points. | 0-8 hours post-dose
  NRS Headache Rating and Characteristics: 0 Minutes (mins) pre-start of GTN, every 15mins to 4 hours (hrs) post-dose, every 30mins to 8hrs post-dose
Pain Response (PR) at 2-hour time point following injection of TRV250 or placebo | every 2 hours for 24 hours
  Two-hour pain response (2HPR; pain response is defined as reduction in migraine type headache severity from verbal NRS score of ≥4 points at 60 minutes post-start of GTN infusion to ≤3 at 24 hours of follow-up)
PF at 2-hour time point following injection of TRV250 or placebo. | every 2 hours for 24 hours
  Two-hour pain freedom (2HPF; pain freedom is defined as reduction in migraine type headache severity from verbal NRS score of ≥4 points at 60 minutes post-start of GTN infusion to ≤1 at 24 hours of follow-up)
Sustained pain response between 2 and 24 hours (2-24H SPR): PR at 2 hours after TRV250 or placebo administration, with no administration of any rescue medication and no occurrence of migraine type headache with verbal NRS score of ≥4 points | up to 24 hours post dose
  Sustained pain response between 2 and 24 hours
Absence of nausea between 2 and 24 hours in patients with nausea from 60 minutes post-start of GTN infusion | up to 24 hours post dose
  Absence of nausea between 2 and 24 hours
Absence of photophobia between 2 and 24 hours in patients with photophobia from 60 minutes post-start of GTN infusion. | up to 24 hours post dose
  Absence of photophobia between 2 and 24 hours
Proportion of patients requiring use of rescue medication at various timepoints. | up to 24 hours of follow-up
  Proportion of patients requiring use of rescue medication at various timepoints.
The effect of TRV250 on cardiac repolarisation determined from cardiac telemetry | Continuous Cardiac Telemetry: min 8hrs pre-GTN to 24hrs post dose
  Patients will be monitored by cardiac telemetry beginning on Day -1 for a minimum of 8 hours pre-GTN infusion and for a minimum of 24 hours post- study drug administration. Any events on cardiac telemetry will be printed and recorded. All cardiac telemetry data will be stored and may be analysed later in the development of TRV250 to evaluate potential drug effects on cardiac conduction and/or as needed to evaluate correlations between cardiac rhythm and symptoms (such as dizziness or palpitations).
The effect of TRV250 on cardiac repolarisation (Cardiac Telemetry) | Continuous Cardiac Telemetry: min 8hrs pre-GTN to 24hrs post dose
  The effect of TRV250 on cardiac repolarisation as determined from cardiac telemetry. Cardiac telemetry will begin on Day -1 a minimum of 8 hours pre-GTN infusion and for 24 hours post-dose. Any events on cardiac telemetry will be printed and recorded. All cardiac telemetry data will be stored and may be analysed later in the development of TRV250 to evaluate potential drug effects on cardiac conduction and/or as needed to evaluate correlations between cardiac rhythm and symptoms (such as dizziness or palpitations).
The effect of TRV250 on cardiac repolarisation (Electrocardiogram) | 12-lead ECG: screening, Day-1 and up to 24 hours post dose
  The effect of TRV250 on cardiac repolarisation as determined from Electrocardiogram (ECG) to check TRV250 effect on the prolongation of QT interval. A 12-lead ECG will be collected at Screening and Day 1 pre-GTN infusion in triplicate, approximately 1 minute apart. ECG will also be collected at single timepoints of: 1-hour, 4-hour and 24-hours post-dose. 12-lead ECGs should be obtained after the patient has rested in the supine position for at least 5 minutes.
Safety Assessment - Injection Site Assessment | at time of GTN-infusion (0 hours) up to 24hrs post-dose
  of pain, tenderness, erythema/redness, and induration/swelling at the injection sites will be conducted pre-GTN infusion, and at 0 hours up to at least 24 hours post-dose.
The PK data model for each patient/dose combination: AUC(0-∞) | up to 24 hours post dose
  AUC from 0 to time infinity (ng∙hr/mL) at Pre-dose, 0.25, btwn 1-3hrs, btwn 6-12hrs, 24hrs
The PK data model for each patient/dose combination: AUC(0-24) | up to 24 hours post dose
  AUC from 0 to 24 hrs post-dose (ng∙hr/mL) at Pre-dose, 0.25, btwn 1-3hrs, btwn 6-12hrs, 24hrs
The PK data model for each patient/dose combination: Cmax (ng/mL) o Tmax - Time of maximum concentration (hours) o t1/2 - half-life (hours) | up to 24 hours post dose
  Cmax (ng/mL) at Pre-dose, 0.25, btwn 1-3hrs, btwn 6-12hrs, 24hrs
The PK data model for each patient/dose combination: Tmax | up to 24 hours post dose
  Time of maximum concentration (hours) at Pre-dose, 0.25, btwn 1-3hrs, btwn 6-12hrs, 24hrs
The PK data model for each patient/dose combination: t1/2 | up to 24 hours post dose
  half-life (hours) at Pre-dose, 0.25, btwn 1-3hrs, btwn 6-12hrs, 24hrs

OTHER OUTCOMES:
Migraine headache relapse defined as a verbal NRS headache score ≥4 points from the timepoint of Pain Response (PR) through 24 hours of follow-up. | up to 24 hours of follow-up
  Migraine headache relapse defined as a verbal NRS headache score ≥4 points from the timepoint of Pain Response (PR) through 24 hours of follow-up.
Sustained pain freedom between 2 and 24 hours (2-24H SPF). | 2-24 hours post dose
  Sustained pain freedom between 2 and 24 hours (2-24H SPF).
Two-hour total migraine freedom (2H TMF; migraine freedom is defined as PF + no nausea + no vomiting + no photophobia + no phonophobia): TMF at 2-hour time point. | 2-hours
  Two-hour total migraine freedom (2H TMF; migraine freedom is defined as PF + no nausea + no vomiting + no photophobia + no phonophobia): TMF at 2-hour time point.
Two-hour total migraine freedom (2H TMF; migraine freedom is defined as PF + no nausea + no vomiting + no photophobia + no phonophobia): TMF at 2-hour time point. | up to 24 hours of follow-up
  Two-hour total migraine freedom (2H TMF; migraine freedom is defined as PF + no nausea + no vomiting + no photophobia + no phonophobia): TMF at 2-hour time point.
Total migraine freedom between 2 and 24 hours (2-24H TMF): 2H + no nausea + no vomiting + no photophobia + no phonophobia between 2 hours and 24 hours after TRV250 or placebo administration. | up to 24 hours of follow-up
  Total migraine freedom between 2 and 24 hours (2-24H TMF): 2H + no nausea + no vomiting + no photophobia + no phonophobia between 2 hours and 24 hours after TRV250 or placebo administration.
Time to pain response (TTPR). | 0-8 hours and up to 24 hours of follow-up
  Time to pain response (TTPR).
Time to pain freedom (TTPF). | 0-8 hours and up to 24 hours of follow-up
  Time to pain freedom (TTPF).
Acute migraine type headache characteristics evoked with GTN infusion compared with spontaneous migraine. | up to 24 hours of follow-up
  Acute migraine type headache characteristics evoked with GTN infusion compared with spontaneous migraine.
Number of evoked headaches that have at least 2 of the 4 migraine characteristic criteria (IHS 1.1 - Criteria C) and have at least 1 of the 2 associated headache criteria (IHS 1.1 - Criteria D). | up to 24 hours of follow-up
  Number of evoked headaches that have at least 2 of the 4 migraine characteristic criteria (IHS 1.1 - Criteria C) and have at least 1 of the 2 associated headache criteria (IHS 1.1 - Criteria D).
Number of evoked headaches that have at least 2 of the 4 migraine characteristic criteria (IHS 1.1 - Criteria C). | up to 24 hours of follow-up
  Number of evoked headaches that have at least 2 of the 4 migraine characteristic criteria (IHS 1.1 - Criteria C).
Number of evoked headaches that have at least 1 of the 2 associated headache criteria (IHS 1.1 - Criteria D). | up to 24 hours of follow-up
  Number of evoked headaches that have at least 1 of the 2 associated headache criteria (IHS 1.1 - Criteria D).
Anxiety monitoring using | up to 24 hours of follow-up
  Change from baseline in Generalised Anxiety Disorder 7-item (GAD-7) Scale at various timepoints post-dose.
Orthostatic assessments - Blood Pressure | at 4 hours post-dose
  Dosing period orthostatic assessments will be measured from Day -30 to Day -2 (pre-dosing) and after the patient stands for 2 minutes (for the first time after dosing). Patients should remain in a supine position, sitting or semi-recumbent for the first 4 hours after dosing
Orthostatic assessments - Heart Rate | at 4 hours post-dose
  Dosing period orthostatic assessments will be measured from Day -30 to Day -2 (pre-dosing) and after the patient stands for 2 minutes (for the first time after dosing). Patients should remain in a supine position, sitting or semi-recumbent for the first 4 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Dasyam, MBBS, Msc, Principal Investigator — MAC Clinical Research Manchester (Early Phase Unit); Nicklas, RN BSN CCRC, Study Director — Trevena Inc.
Locations (1):
- MAC Clinical Research Manchester (Early Phase Unit), Neuroscience Centre of Excellence, Manchester, Greater Mancherster, United Kingdom

IPD SHARING:
Plan to Share IPD: No